CLINICAL TRIAL: NCT00197691
Title: Botswana Pediatric Respiratory Disease and Bloodstream Infection
Brief Title: Botswana Pediatric Respiratory Disease and Bloodstream Infection Study
Status: Completed | Type: Observational
Sponsor: Harvard School of Public Health (HSPH) (Other)
Responsible Party: Sponsor
Other Study IDs: HSC 10027/000BOTS
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2012-04-02 (Estimated); Status verified 2012-03

CONDITIONS: HIV Infections; Respiratory Tract Diseases; Sepsis
Keywords: HIV infected mothers; Infants at risk of HIV-infection; Infant lower respiratory tract disease; Infant bloodstream infection
MeSH Terms: conditions — HIV Infections; Respiratory Tract Diseases; Sepsis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: blood draws, etc.

SUMMARY:
The purpose of this study is to learn about lower respiratory tract and bloodstream diseases among infants born to HIV positive mothers in Botswana. Study factors include how commonly infants get these diseases, the causes, and outcomes. The study will also try to measure the protective effect, if any, of breast feeding on respiratory disease illness and deaths.

ELIGIBILITY:
Inclusion Criteria:

* Participation in parent study, "Mashi" HIV vertical transmission prevention study for pregnant Botswana women and their infants

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: LIVEBORN INFANT IN THE MASHI PMTCT TRIAL
Sampling Method: Non-Probability Sample
Dates: Start 2001-03; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
OCCURRENCE OF SUSPECTED PNEUMONIA OR BLOODSTREAM INFECTION OVER FIRST TWO YEARS OF LIFE | Between birth and 2 years of life
  MORTALITY; EPISODES OF SUSPECTED PNEUMONIA; BACTEREMIA; PRESENCE OF NASOPHARYNGEAL VIRAL PATHOGENS; OROPHARYNGEAL COLONIZATION WITH BACTERIAL PATHOGENS

CONTACTS AND LOCATIONS:
Overall Officials: Shahin Lockman, MD, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- Princess Marina Hospital, Gaborone, Botswana

REFERENCES:
- [Derived] Shapiro RL, Smeaton L, Lockman S, Thior I, Rossenkhan R, Wester C, Stevens L, Moffat C, Arimi P, Ndase P, Asmelash A, Leidner J, Novitsky V, Makhema J, Essex M. Risk factors for early and late transmission of HIV via breast-feeding among infants born to HIV-infected women in a randomized clinical trial in Botswana. J Infect Dis. 2009 Feb 1;199(3):414-8. doi: 10.1086/596034. PMID 19090775
- [Derived] Shapiro RL, Lockman S, Kim S, Smeaton L, Rahkola JT, Thior I, Wester C, Moffat C, Arimi P, Ndase P, Asmelash A, Stevens L, Montano M, Makhema J, Essex M, Janoff EN. Infant morbidity, mortality, and breast milk immunologic profiles among breast-feeding HIV-infected and HIV-uninfected women in Botswana. J Infect Dis. 2007 Aug 15;196(4):562-9. doi: 10.1086/519847. Epub 2007 Jul 9. PMID 17624842